CLINICAL TRIAL: NCT06370962
Title: Overview of Circadian Rhythm Disorders in Children With Cystic Fibrosis in the Era of CFTR (Cystic Fibrosis Transmembrane Conductance Regulator) Modulators
Brief Title: Circadian Rhythm Disorders in Children With Cystic Fibrosis Under CFTR (Cystic Fibrosis Transmembrane Conductance Regulator) Modulators
Acronym: CHRONO-MUCO
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0076; 2024-A00343-44 (Other: ID-RCB)
Record Dates: First submitted 2024-02-19; First posted 2024-04-17 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; Cystic fibrosis transmembrane conductance regulator modulators; circadian rhythm disorders
MeSH Terms: conditions — Cystic Fibrosis; Chronobiology Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of urine samples for urinary melatonin determination will be carried out only for patients in the Lyon group for technical reasons (sleep disorders reference laboratory in Lyon; not available in Paris and Nancy).
  These samples will only be collected in Lyon patients with sleep complaints, as they are specific to the current care practice in Lyon.
  4 tubes of around 10 ml will be collected per patient. Urine samples will be analyzed at the Lyon Hormone Analysis Laboratory - Louis Pradel Hospital (Dr Véronique Raverot, reference medical biology laboratory for sleep pathologies). Analysis will be carried out during the course of the study as samples arriving, in accordance with the department's standard practice.
  Urine samples will be traced from collection to the laboratory. All samples will be used for analysis; samples will not be stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adolescents with cystic fibrosis treated with Kaftrio-Kalydeco: Patients with cystic fibrosis Aged from 2 to 17 years and 11 months Treated with CFTR modulator Kaftrio-Kalydeco for at least 2 months Followed in a participating Cystic Fibrosis Resource and Skill national Centre

SUMMARY:
Cystic fibrosis (CF) is a rare disease affecting one out of 4,500 newborns in France (INSERM 2021). Despite major advances in patient care over the past two decades, with significant improvements in life expectancy, cystic fibrosis remains a pathology that considerably impairs quality of life.

Several studies have reported the possibility of respiratory and non-respiratory sleep disorders (SD) in patients with CF. Respiratory disorders are reported to affect 30% of children with CF (Barbosa 2020). Among non-respiratory SD, sleep onset and maintenance insomnia are well known in these patients, while chronotype abnormalities (circadian rhythm disorders) are understudied. Chronotype refers to a person's tendency to be more efficient in the morning or evening.

The existence of chronotype abnormalities has been suggested in CF patients, but no precise data are available (Louis 2022). The involvement of CFTR (Cystic Fibrosis Transmembrane Conductance Regulator) protein dysfunction in the central nervous system (CNS) has been hypothesized as a contributory factor. In vivo, in a mouse model of CF, dysregulation of clock genes such as Clock, Cry2 and Per2 was found in the CNS (Barbato 2019). Among them, certain genes such as Rev-erbα could regulate endobronchial inflammation and contribute to the severity of respiratory pathology. All in all, chronotype abnormalities could be at the origin of sleep debt, impaired cognitive functions or metabolic disturbances.

In the era of highly effective modulator therapy (HEMT) for the treatment of CF, the impact of these new therapies on chronotype has been understudied. Assuming that chronotype abnormalities are a direct consequence of CFTR protein dysfunction in the retina and anterior hypothalamus, HEMT should improve sleep quality. However, between 20% and 30% of adult and pediatric patients express an increase in chronotype abnormalities following initiation of treatment.

Paradoxically, the perceived gain in respiratory quality of life is counterbalanced by the occurrence of these disorders. Some patients would effectively reverse their treatment in order to limit the phenomenon. A single polysomnographic study evaluated the effect of HEMT Kaftrio-Kalydeco on sleep in adults with CF (Welsner 2022). After 3 months of treatment, patients had a significant reduction in respiratory events, with no change in total sleep time, sleep efficiency or sleep architecture. Chronotype was not mentioned. Currently, no studies on chronotype in children or adults with CF have been carried out. Our hypothesis is that CF patients treated with HEMT would develop an abnormal chronotype of late sleep onset.

The aim of this study is to evaluate the chronotype of children with CF treated with HEMT. Chronotype abnormalities could have major consequences for quality of life, the immune system, cognitive functions and metabolism. Systematic detection of these disorders via anamnesis, followed by diagnosis by questionnaire, actimetrics and/or urinary melatonin dosage, would enable their early management, starting with the reversal of Kaftrio-Kalydeco intake between morning and evening.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cystic fibrosis
* Aged from 2 to 17 years and 11 months
* Treated with CFTR modulator Kaftrio-Kalydeco from at least 2 months
* Followed in Lyon, Paris-Trousseau or Nancy Cystic Fibrosis Resource and Skill Centres
* Non-opposition from both parents

Exclusion Criteria:

* Parental refusal
* Parents unable to comply with protocol requirements at investigator's discretion
* Subject participating in interventional research with an exclusion period still in progress at the time of inclusion

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will be selected from Cystic Fibrosis Resource and Skill Centres of pediatric tertiary care hospitals (Lyon, Paris-Trousseau, Nancy).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-10-29 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Result of the Horne and Ostberg questionnaire. | Day 0
  The frequency of each chronotype (normal, morning or evening) in patients with CF on HEMT will be determined by the result of the Horne and Ostberg questionnaire.
  The frequency of each chronotype will be summarized for all CF patients on HEMT using the following descriptive statistics: frequencies and percentages for each level of the variable (normal, morning or evening) and the number of missing values (missing values will be counted but not included in the denominator of the frequency calculation).
  Scores from 5 to 25: 21-25 = clearly morning; 18-20 = moderately morning; 12-17 = nor morning, neither evening; 9-11: moderately evening; 5-8: clearly evening.

CONTACTS AND LOCATIONS:
Overall Officials: Laurianne COUTIER, MD, Principal Investigator — Service de pneumologie, allergologie, mucoviscidose, Hôpital Femme Mère Enfant, HCL
Locations (3):
- France (3):
  - Hôpital Femme Mère Enfant, Bron
  - Service de pédiatrie, CHRU de Nancy - Hôpitaux de Brabois, Nancy
  - Service de pneumologie pédiatrique, Hôpital Armand Trousseau, Paris